CLINICAL TRIAL: NCT03104946
Title: Clinical Research on the Predictive Effect of Neonatal Morbidities on the Poor Outcomes to Very Low Birth-weight and Extremely Low Birth-weight Infants
Brief Title: To Research the Relation Between Neonatal Morbidities and Poor Outcome in Preterm Infants
Status: Completed | Type: Observational
Sponsor: yangjie (Other)
Responsible Party: Sponsor-Investigator, yangjie, Director of Dept of Neonatology, Guangdong Women and Children Hospital
Organization: Guangdong Women and Children Hospital (Other)
Other Study IDs: Guangdong WCH
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Preterm Infant; Morbidity;Infant; Outcome, Fatal
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Bronchopulmonary Dysplasia
  Interventions: Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus
- Retinopathy
  Interventions: Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus
- Severe Retinopathy
  Interventions: Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus
- Neonatal Necrotizing Enterocolitis
  Interventions: Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus
- Brain injury
  Interventions: Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus
- sepsis
  Interventions: Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus
- Patent Ductus Arteriosus
  Interventions: Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus
- Respiratory Distress Syndrome
  Interventions: Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus

INTERVENTIONS:
Diagnostic Test: Mental Development Index;Auditory Brainstem Response;okineticnystagmus — mental development index(MDI）<70:cognitive delay do not pass auditory brainstem response(ABR）：hearing impairment do not pass okineticnystagmus:visual impairment Patent Ductus Arteriosus

SUMMARY:
From November 2014 to October 2015, a multi-centers retrospective study was conducted to collect compliance, and 8 three-level hospitals from China were included. The infants survived to a postmenstrual age of 36 week with birth weight less than 1500g and without congenital disease. The birth weight, gestational age, morbidities and poor outcomes( death, cerebral palsy, cognitive, et al) were recorded. Data were analyzed with Chi-square test to observe the relationship between morbidities and poor outcomes. And the predictive effect on the number of the top three morbidities were analyzed by Logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

From November 2014 to October 2015, a multi-centers retrospective study was conducted to collect compliance, and 8 three-level hospitals from China were included. The infants survived to a postmenstrual age of 36 week with birth weight less than 1500g.

Exclusion Criteria:

The very low birth weight infants didn't have any congenital disease.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: From November 2014 to October 2015, a multi-centers retrospective study was conducted to collect compliance, and 8 three-level hospitals from China were included. The infants survived to a postmenstrual age of 36 week with birth weight less than 1500g and without congenital disease.
Sampling Method: Non-Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
cognitive delay | 1 year
  mental development index(MDI）<70
hearing impairment | 1 year
  do not pass auditory brainstem response (ABR)
visual impairment | 1 year
  do not pass okineticnystagmus

REFERENCES:
- [Background] Schmidt B, Asztalos EV, Roberts RS, Robertson CM, Sauve RS, Whitfield MF; Trial of Indomethacin Prophylaxis in Preterms (TIPP) Investigators. Impact of bronchopulmonary dysplasia, brain injury, and severe retinopathy on the outcome of extremely low-birth-weight infants at 18 months: results from the trial of indomethacin prophylaxis in preterms. JAMA. 2003 Mar 5;289(9):1124-9. doi: 10.1001/jama.289.9.1124. PMID 12622582
- [Derived] Rao YB, Yang J, Cao B, Chen DM, Gao PM, Zhong Q, Li MX, Gao JH, Chen YJ, Zhong XM, Ren ZX. [Predictive effect of neonatal morbidities on the poor outcomes at 12 months corrected age in very low birth weight premature infants]. Zhonghua Er Ke Za Zhi. 2017 Aug 2;55(8):608-612. doi: 10.3760/cma.j.issn.0578-1310.2017.08.012. Chinese. PMID 28822437